CLINICAL TRIAL: NCT01620385
Title: Multi Center Clinical Study to Assess the Safety of the UTD Cochlear Implant PDA (ciPDA) REsearch Platform
Brief Title: Cochlear Implant PDA Based Research Platform
Acronym: ciPDA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philip Loizou (Other)
Responsible Party: Sponsor-Investigator, Philip Loizou, PI, The University of Texas at Dallas
Organization: The University of Texas at Dallas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ciPDA0001
Record Dates: First submitted 2011-09-08; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Hearing Impaired
Keywords: Cochlear implants
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ciPDA (Experimental)
  Interventions: Device: ciPDA

INTERVENTIONS:
Device: ciPDA — The ciPDA Research Platform device was designed as a research tool for cochlear implant research.
  Other Names: Single arm study.

SUMMARY:
The primary purpose of the research is to study how individuals who wear cochlear implants process sounds in noisy environments and also whether newly designed programs can help improve the communicative ability of cochlear implant patients in noisy situations.

DETAILED DESCRIPTION:
Cochlear implants have been successful in restoring partial hearing to profoundly deaf people. Despite their success, most implant patients are not able to communicate in noisy environments (e.g., in a restaurant). Communicating in noise still remains one of the biggest challenges in cochlear implants. Little is known about the factors that contribute to the poor performance of CI users in noise. In this project, we propose a series of experiments aimed at isolating these factors. We propose new programs that can be tailored for noisy situations.

ELIGIBILITY:
Inclusion Criteria:

1. Post-lingually deafened adults:

   * 18 years of age or older
   * Unilateral or bilateral Nucleus implant users (this includes all three generations of the Nucleus system, i.e., CI22, CI24 and CI24R).
   * With or without residual hearing in the contralateral ear. Subjects may use amplification (hearing aid) in the opposite or same ear as the implant.
   * A minimum test score of 30% in tape-recorded open-set sentence recognition scores (e.g., spondee identification).
   * Minimum of 6 months experience with their implant device. This is done to ensure that all patients are familiar with the hearing sensations perceived by a cochlear implant.
   * Minimum number of active electrodes: 10
   * Minimum number of subjects for each test site: 5
2. Prelingually and perilingually deafened adults:

   * 18 years of age or older
   * Unilateral or bilateral Nucleus implant users.
   * With or without residual hearing in the contralateral ear. Subjects may use amplification (hearing aid) in the opposite or same ear as the implant.
   * A minimum test score of 10% in tape-recorded open-set sentence recognition scores (e.g., spondee identification).
   * Minimum of 6 months experience with their implant device. This is done to ensure that all patients are familiar with the hearing sensations perceived by a cochlear implant.
   * Minimum number of active electrodes: 10
   * Minimum number of subjects for each test site: 5

Exclusion Criteria:

* Non-English speaking
* Hearing loss of neural or central origin
* Absence of cochlear or VIII nerve development
* The presence of systemic condition which would preclude use of a cochlear implant
* Active middle ear infection/tympanic membrane perforation
* Significantly abnormal cognitive function, as determined by case history information and/or clinical observations
* Significant psychiatric disorder, as determined by case history information and/or clinical observations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The objective of this study is to assess the safety of the PDA device after long-term use. Safety shall be measured by the adverse events reported in this study and compared to the study results reported in the clinical study for the PMA'd device. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Loizou, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas - Dallas, Richardson, Texas, United States